CLINICAL TRIAL: NCT06756555
Title: Effect of Incentive Spirometry on Post Operative Pulmonary Complications After Bariatric Surgery: a Cross Sectional Study
Brief Title: Effect of Incentive Spirometry on Post-operative Pulmonary Complications After Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/019
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: efficacy of Incentive spirometer — The main objective of this research is to check the efficacy of Incentive spirometer on pulmonary complication after bariatric surgrey

SUMMARY:
Today, obesity is the major concern and obese patients are at higher risk of developing pulmonary complications. Incentive Spirometry is widely used worldwide to reduce rates of pulmonary complications. In this study, Effect of Incentive Spirometry (IS) on Post Operative Bariatric Patients (Male and Female) will be studied on patients about sample size of 140 including male and female gender, BMI above 30 kg/m2 having Post Operative Bariatric Surgeries with chances of generating Pulmonary complications.

DETAILED DESCRIPTION:
Research will be conducted in Shalamar Hospital Lahore and data will be collected through predesigned proforma. In previous studies some studies show positive and but some studies don't recommend Incentive Spirometry as a post operative Rehabilitation therapy.But this therapy device is still used in present days in Post Operative patients to prevent pulmonary complications. In this study we conclude the positive or negative effect of Incentive Spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Patient having weight above 25 BMI
* Age between 18 years to 60 years
* having Post Operative pulmonary complication.
* Bariatric patients (Sleeve gastrectomy,Mini gastric Bypass,Sleeve gastrectomy to gastric bypass ,sleeve re do surgery)..

Exclusion Criteria:

* Patients weight below 25BMI.
* other abdominal surgeries.
* Patients having absence of teeth.
* Patients age below 18 years .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: population included Complications After Bariatric Surgery to check the Effects of Incentive Spirometry on Post-operative Pulmonary
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate using Spirometry | 12 Months
  Rrespiratory rate, assessed using manual or electronic monitoring, and patient satisfaction with incentive spirometry, evaluated through a structured questionnaire focusing on ease of use and perceived benefits.
  Average values in healthy patients aged 20-60 range from 5.5 to 4.75 liters in males and from 3.75 to 3.25 liters in females.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital Mughalpura, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No